CLINICAL TRIAL: NCT00572117
Title: Adjunctive Topiramate for Treatment of Alcohol Dependence in Patients With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Michael Ostacher, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TIL-NIAAA-016340-01; K23AA016340 (NIH)
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Bipolar Disorder; Alcoholism; Alcohol Dependence
Keywords: Bipolar Disorder; Manic Disorder; Alcoholism; Alcohol Abuse; Alcohol Dependence; Clinical Trial; Evaluation Trial; Intervention Trial; Validation Studies
MeSH Terms: conditions — Bipolar Disorder; Alcoholism | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (inert pill) Arm (Placebo Comparator): Half the participants will receive topiramate and half will receive placebo. Neither participants nor study staff will know who is receiving which pills until the end of the study. Subjects will receive placebo pills identical to the active pills (pills that contain the study drug, topiramate) for the 12 treatment weeks of the study and will have the pills discontinued over the next four weeks of the study. All subjects will be re-evaluated at 26 and 52 weeks.
  Interventions: Drug: Topiramate
- Topiramate (Experimental): Half the participants will receive topiramate and half will receive placebo. Neither participants nor study staff will know who is receiving which pills until the end of the study. The pills will be slowly increased over 5 weeks from 25 mg a day to 150 mg twice a day in an effort to minimize side effects that might enable participants and raters to guess whether they are on active drug or placebo. Subjects will continue on 150 mg twice a for Weeks 6-12 of the study.
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Medication will be slowly increased over 5 weeks from 25 mg a day to 150 mg twice a day in an effort to minimize side effects that might enable participants and raters to guess whether they are on active drug or placebo. Subjects will continue on 150 mg twice a for Weeks 6-12 of the study.
  Other Names: Topamax

SUMMARY:
The purpose of this study is determine whether the use of topiramate is effective in the treatment of alcohol dependence (i.e. decreases drinking) in patients with bipolar disorder.

DETAILED DESCRIPTION:
Alcohol and substance use disorders are more common in bipolar disorder bipolar disorder than in any other DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) Axis I disorder, estimated to occur in up to 60% of patients with bipolar disorder. Alcohol use is associated with poor outcome in bipolar disorder, and yet these co-occurring conditions are understudied. To date, there is only one published placebo-controlled trial of an agent for the treatment of alcohol dependence alcohol dependence in bipolar disorder. The purpose of the proposed study is to evaluate the efficacy of a topiramate as a treatment for alcohol dependence in patients with bipolar disorder. This is a 12-week, randomized, placebo-controlled study of the efficacy of topiramate adjunctive to standard treatment for bipolar disorder in patients with alcohol dependence and bipolar disorder. Additional aims of the study are to document the safety and tolerability of topiramate in this population, and to evaluate to effect of decreased drinking on mood symptoms. The study involves the enrollment of a total of 80 patients with co-occurring alcohol dependence and bipolar disorder over the course of 40 months at the Massachusetts General Hospital (MGH) Bipolar Clinic and Research Program (BCRP) (www.manicdepressive.org). With a conservative estimate of a 30% dropout rate, approximately 56 of the 80 patients with these two comorbid conditions will complete 12 weeks treatment with either topiramate or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. Written informed consent.
3. Meet DSM-IV criteria (by SCID) for alcohol dependence.
4. Meet DSM-IV criteria (by SCID) for bipolar disorder I or II disorder.
5. ≥ 8 heavy drinking days (defined as ≥ 5 standard drinks per day for men, ≥ 4 standard drinks per day for women) in the prior 4 weeks.
6. During the baseline visit, patients must be on a stable dose of accepted maintenance treatment for bipolar disorder for the past 4 weeks. If the subject is on more than one agent, at least one agent must be adequately dosed.
7. Antidepressant treatment is permitted if the dose has been stable for the past 4 weeks.

Exclusion Criteria:

1. Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy). Because of the risk of the lowering of oral contraceptive blood levels with topiramate, women whose sole means of contraception is oral contraceptives or hormonal implants will be asked to use an additional barrier method of birth control during treatment with the study drug.
2. Women who are lactating.
3. Age under 18.
4. Patients who do not have ≥ 8 heavy drinking days in the 4 weeks prior to the baseline visit.
5. Important alcohol withdrawal symptoms (Clinical Institute Withdrawal Assessment for Alcohol-Revised, CIWA-Ar, score > 15)
6. Urine toxicological screen positive for amphetamines or cocaine.
7. Meets DSM-IV criteria for current substance dependence for drugs other than cannabis or nicotine.
8. Currently meets full DSM-IV criteria for manic, hypomanic, or mixed episode.
9. Serious suicide or homicide risk, as assessed by evaluating clinician.
10. Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease or uncontrolled seizure disorder.
11. History of nephrolithiasis, or treatment with any drug associated with nephrolithiasis.
12. Current treatment with zonisamide.
13. Current treatment with any carbonic anhydrase inhibitors, including acetazolamide, dorzolamide, and methazolamide.
14. Current treatment with any drug known to decrease drinking.
15. Subjects who have begun a new psychosocial treatment within 12 weeks of study enrollment. Subjects receiving psychosocial treatment that has been stable for at least 12 weeks prior to study entry, however, will be permitted to enroll in the study.
16. Any psychotic disorder, including schizoaffective disorder (current or past).
17. Clinical or laboratory evidence of untreated hypothyroidism.
18. Patients with a diagnosis or history of glaucoma
19. Patients requiring excluded medications (see table below for details).
20. Psychotic features in the current episode or a history of a psychotic disorder, as assessed by SCID.
21. Past intolerance to topiramate.
22. Any use of topiramate in the past 12 months.
23. Any investigational psychotropic drug within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Ostacher, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Stanford/VA Palo Alto Mood Disorder Research Program, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topiramate | Placebo (Inert Pill) Arm
Started | 5 | 7
Completed | 3 | 5
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo (Inert Pill) Arm | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (10.8) | 46.6 (8.3) | 43.6 (9.7)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Amount of Alcohol Consumed
Description: Average number of drinks/heavy drinking days/week as measured using the Timeline Follow Back (TLFB) scale. A heavy drinking day is defined as a 5 or more standard drinks in a single day for males, 4 or more standard drinks in a single day for females. Drinks are standardized across types of alcohol to estimate the amount of alcohol consumes. For example, a 12 oz. beer of 4-5% alcohol by volume is considered one drink.
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: number of drinks per heavy drinking day
Groups:
- Topiramate; Placebo (Inert Pill) Arm: Change in average number of drinks/heavy drinking day
Arm/Group | Topiramate | Placebo (Inert Pill) Arm
Number analyzed (Participants) | 5 | 7
number of drinks per heavy drinking day | -1.38 [-4.93 to 2.17] | -0.69 [-1.68 to 0.31]

2. Secondary Outcome: Effect of Treatment on Mood Symptoms
Description: The 17-item Hamilton Depression Rating Scale (HAM-D) is a standard measure of symptoms of depression with a scoring range of 0-53 points. Higher HAM-D scores represent more depression, so a lowering of HAM-D scores is considered a good outcome, an increase in HAM-D scores considered a worsening of outcomes.
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Topiramate; Placebo (Inert Pill) Arm: Change in HAM-D score from baseline
Arm/Group | Topiramate | Placebo (Inert Pill) Arm
Number analyzed (Participants) | 5 | 7
units on a scale | -2.00 [-6.21 to 2.21] | -0.72 [-8.96 to 7.54]

ADVERSE EVENTS:
Arm/Group | Topiramate | Placebo (Inert Pill) Arm
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/7
Other Adverse Events (participants affected / at risk) | 1/5 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=5) | Placebo (Inert Pill) Arm (N=7)
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=5) | Placebo (Inert Pill) Arm (N=7)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No